CLINICAL TRIAL: NCT07345832
Title: Digital Pathway to Healthy Aging: Sarcopenia-Frailty Integrated Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-Path-HA: S-FIT
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Sarcopenia in Elderly; Fall Prevention in Healthy Aging; Frailty; Malnutrition Elderly
Keywords: sarcopenia; elderly; frailty; fall prevention; malnutrition; health-related quality of life; digital intervention
MeSH Terms: conditions — Sarcopenia; Frailty; Malnutrition

STUDY DESIGN:
Intervention Model Description: This Randomized Controlled Trial randomized 200 older adults with risk of, or diagnosed with, sarcopenia and frailty to receive the digital pathway intervention or a waiting list control group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the intervention assignment results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Pathway to Healthy Aging: Sarcopenia-Frailty Integrated Training program (Experimental): This digital program will address sarcopenia and frailty with a 12-week integrated intervention based on integrated exercise, nutrition, and fall-prevention.
  Interventions: Behavioral: Digital Pathway to Healthy Aging: Sarcopenia-Frailty Integrated Training program (D-Path-HA: S-FIT)
- Waitlist Control (Active Comparator): The control group will receive general education on nutrition and physical activity guidelines for older adults, and the same pathway intervention will be applied to the control group after all data collection
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Digital Pathway to Healthy Aging: Sarcopenia-Frailty Integrated Training program (D-Path-HA: S-FIT) — This digital program will address sarcopenia and frailty with a 12-week integrated intervention based on integrated exercise, nutrition, and fall-prevention. The intervention will be delivered by registered nurses, social workers, and health coach captains. Guided by the critical pathway and empowerment cycle framework, including a (1) Personalised Health Prescription Phase, (2) 12-Week Empowerment and Social Activity Phase, including six bi-weekly, in-person sessions empowerment workshop; scenario-based health message broadcast; case meeting.
  Arms: Digital Pathway to Healthy Aging: Sarcopenia-Frailty Integrated Training program
Behavioral: Waitlist Control — The control group will receive general education on nutrition and physical activity guidelines for older adults, and the same pathway intervention will be applied to the control group after all data collection.
  Arms: Waitlist Control

SUMMARY:
Sarcopenia and frailty prevention and management are highly prioritized goals in the Healthy Aging agenda. The study aims to evaluate the effects and implementation of the digital critical pathway to improve sarcopenia and frailty, reduce fall risk, and increase health-related quality of life among community-dwelling older adults with risk of, or diagnosed with, sarcopenia and frailty

DETAILED DESCRIPTION:
Population ageing is accelerating globally and regionally, widening the gap between life expectancy and healthy life expectancy, mainly due to late-life declines in physical function and mobility (Guo et al., 2022). Sarcopenia and frailty are major age-associated public health issues that contribute to a decline in functional ability, increased fall risks, and mortality (Lee et al., 2022; Petermann-Rocha et al., 2021). Nutrition and physical activity integrated interventions are recommended as primary treatment for sarcopenia and frailty (Park & Lee, 2023). However, current interventions are often generic, resulting in non-precise, non-personalized interventions, usually failing to accommodate individual differences in baseline strength and mobility, nutrition status, comorbidities, preferences, and home environments (Tighe et al., 2020). Consequently, interventions are complex to personalise, adjustments are delayed, and adherence is suboptimal, undermining real-world effectiveness. Future community-based health agendas should prioritize long-term care that removes access barriers (such as mobility and transportation) and transitions from generic care to precision personalization.

The World Health Organisation's Decade of Healthy Ageing and the Integrated Care for Older People (ICOPE) framework provide a practice anchor to maintain intrinsic capacity through person-centred assessment, individualised goal-setting, and continuous follow-up. Within this paradigm, sarcopenia and frailty management apply ICOPE via protocol-driven critical pathways (Sum et al., 2022)-structured decision support that links risk assessment to tailored prescriptions and follow-up-can standardise quality while enabling precise personalisation across diverse home settings.

Digital health interventions have expanded their capabilities to include remote exercise prescription, microlearning, reminders, and tele-coaching, with evidence of benefits for physical activity, fitness, body composition, and patient-reported outcomes (De Santis et al., 2023). Utilising a user-friendly digital tool to streamline functional assessments and develop personalised health plans is a promising approach.

A digital platform-enabled intervention, grounded in the WHO ICOPE framework and a protocol-driven critical pathway, is proposed to identify care needs among community-dwelling older adults. This tool will allow healthcare providers to accurately assess individual needs and tailor interventions in exercise and nutrition, ensuring a focused, effective approach to combating sarcopenia and frailty in older adults.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* Pseudo-Sarcopenia/Sarcopenia: SARC-CaIF ≥ 11, AND (Grip Strength on dominant hand (male <28 kg, female <18 kg), OR Chair Stand Test (5 times) ≥ 12 seconds, OR Short Physical Performance Battery Score ≤ 9; OR relative appendicular skeletal mass/ height (Men: <7 kg/m2; women: <5.7 kg/m2) ); AND/OR Prefrail/ frail based on the Edmonton Frail Scale Score ≥ 6.
* consent to participate

Exclusion Criteria:

* having conditions contradictory to physical activity
* engaging in other ongoing physical activity and nutrition programs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass index (ASMI) | Baseline (T0), 3 months (T1), and 6 months (T2)
  Appendicular skeletal muscle mass index (ASMI) measured by Bioelectrical impedance analysis (BIA)
Handgrip Strength | Baseline (T0), 3 months (T1), and 6 months (T2)
  Handgrip strength will be measured by a hydraulic hand dynamometer from dominant hand, taking the highest value among 3 measurements. Low muscle strength is defined if male <28kg, and femal <18kg.
Short Physical Performance Battery (SPPB) | baseline (T0), 3 months (T1), and 3 months (T2)
  Physical function will be measured by the Short Physical Performance Battery (SPPB), which combines balance test, gait velocity and chair stand. SPPB score ranges from 0-12, higher score better physical performance. Low physical function is defined by SPPB score ≤9.

SECONDARY OUTCOMES:
Sarcopenia and calf circumference scale (SARC-CalF) | Baseline (T0), 3 months (T1), and 6 months (T2)
  Sarcopenia and calf circumference scale (SARC-CalF) includes 5 items (strength, assistance with walking, rising from a chair, climbing stairs, Falls, calf circumference). The score ranges from 0 to 20 points, with a score ≥ 11 points suggestive of sarcopenia.
11-item Edmonton Frail Scale | Baseline (T0), 3 months (T1), and 6 months (T2)
  The Edmonton Frail Scale (EFS) is scored from 0 to 17, with higher scores indicating greater frailty. An EFS score ≥ 8 is generally used as the cutoff for frailty. Scores 6-7 flag patients who are at risk.
Timed Up and Go (TUG) test | Baseline (T0), 3 months (T1), and 6 months (T2)
  Measured by the Timed Up and Go Test in unit of second. A shorter completion time indicates better mobility and balance.
The Mini Nutritional Assessment (MNA) | Baseline (T0), 3 months (T1), and 6 months (T2)
  Measured by the Mini Nutritional Assessment (scores range from 0 to 30), with a lower score indicating a higher risk of malnutrition.
International Physical Activity Questionnaire (IPAQ-Short) | Baseline (T0), 3 months (T1), and 6 months (T2)
  Measured by International Physical Activity Questionnaire is a self-report measure of physical activity. Frenquency and time spent on walking, moderate and vigorous physical activity will be reported. More time spent on physical actiivty indicating a higher physical activity level.
Sleep duration | Baseline (T0), 3 months (T1), and 6 months (T2)
  Sleep duration in daytime and night on weekday and weekend
The EuroQoL-5D-5L instruments | Baseline (T0), 3 months (T1), and 6 months (T2)
  Assess the health-related quality of life to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems , moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang Y, Pan N, Luo J, Liu Y, Ossowski Z. Exercise and Nutrition for Sarcopenia: A Systematic Review and Meta-Analysis with Subgroup Analysis by Population Characteristics. Nutrients. 2025 Jul 17;17(14):2342. doi: 10.3390/nu17142342. PMID 40732966
- [Result] Wu S, Nan J, Chang J, Jiang D, Cao Z, Zhou S, Feng H, Xiao LD. Adherence to exercise intervention for community-dwelling older adults with sarcopenia: a systematic review and meta-analysis. Age Ageing. 2025 Mar 28;54(4):afaf094. doi: 10.1093/ageing/afaf094. PMID 40253683
- [Result] Wang Z, Xu X, Gao S, Wu C, Song Q, Shi Z, Su J, Zang J. Effects of Internet-Based Nutrition and Exercise Interventions on the Prevention and Treatment of Sarcopenia in the Elderly. Nutrients. 2022 Jun 14;14(12):2458. doi: 10.3390/nu14122458. PMID 35745187
- [Result] Vijayananthan A, Nawawi O. The importance of Good Clinical Practice guidelines and its role in clinical trials. Biomed Imaging Interv J. 2008 Jan;4(1):e5. doi: 10.2349/biij.4.1.e5. Epub 2008 Jan 1. PMID 21614316
- [Result] Tighe SA, Ball K, Kensing F, Kayser L, Rawstorn JC, Maddison R. Toward a Digital Platform for the Self-Management of Noncommunicable Disease: Systematic Review of Platform-Like Interventions. J Med Internet Res. 2020 Oct 28;22(10):e16774. doi: 10.2196/16774. PMID 33112239
- [Result] Sum G, Lau LK, Jabbar KA, Lun P, George PP, Munro YL, Ding YY. The World Health Organization (WHO) Integrated Care for Older People (ICOPE) Framework: A Narrative Review on Its Adoption Worldwide and Lessons Learnt. Int J Environ Res Public Health. 2022 Dec 22;20(1):154. doi: 10.3390/ijerph20010154. PMID 36612480
- [Result] Rodrigues B, Judice PB, Marques A, Carraca EV, Lopes L, Sousa-Sa E, Encantado J, Videira-Silva A, Cliff DP, Mendes R, Santos R; QMov24h working group. 24-hour Movement Questionnaire (QMov24h) for adults: development process and measurement properties. Int J Behav Nutr Phys Act. 2024 Oct 9;21(1):116. doi: 10.1186/s12966-024-01667-7. PMID 39385225
- [Result] Petermann-Rocha F, Gray SR, Pell JP, Ho FK, Celis-Morales C. The joint association of sarcopenia and frailty with incidence and mortality health outcomes: A prospective study. Clin Nutr. 2021 Apr;40(4):2427-2434. doi: 10.1016/j.clnu.2020.10.044. Epub 2020 Nov 1. PMID 33189425
- [Result] Perna S, Francis MD, Bologna C, Moncaglieri F, Riva A, Morazzoni P, Allegrini P, Isu A, Vigo B, Guerriero F, Rondanelli M. Performance of Edmonton Frail Scale on frailty assessment: its association with multi-dimensional geriatric conditions assessed with specific screening tools. BMC Geriatr. 2017 Jan 4;17(1):2. doi: 10.1186/s12877-016-0382-3. PMID 28049443
- [Result] Pek K, Tan CN, Yew S, Yeo A, Lim JP, Chew J, Lim WS. Letter to the Editor: COVID-19 Pandemic Control Measures: Impact on Social Frailty and Health Outcomes in Non-Frail Community-Dwelling Older Adults. J Nutr Health Aging. 2021;25(6):816-818. doi: 10.1007/s12603-021-1635-1. No abstract available. PMID 34179939
- [Result] Park SH, Lee H. Effectiveness of Combined Exercise and Nutrition Interventions in Preventing and Improving Sarcopenia in Frail or Healthy Older Adults: A Systematic Review. Res Gerontol Nurs. 2023 Nov-Dec;16(6):312-320. doi: 10.3928/19404921-20230817-03. Epub 2023 Aug 25. PMID 37616483
- [Result] Meza-Valderrama D, Sanchez-Rodriguez D, Pena YC, Ramirez-Fuentes C, Munoz-Redondo E, Morgado-Perez A, Ortiz-Agurto N, Finis-Gallardo P, Marco E. Resistance Training and Nutritional Supplementation in Older Adults with Sarcopenia after Acute Disease: A Feasibility Study. Nutrients. 2024 Sep 10;16(18):3053. doi: 10.3390/nu16183053. PMID 39339653
- [Result] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Result] Lee D, Kim M, Won CW. Common and different characteristics among combinations of physical frailty and sarcopenia in community-dwelling older adults: The Korean Frailty and Aging Cohort Study. Geriatr Gerontol Int. 2022 Jan;22(1):42-49. doi: 10.1111/ggi.14314. Epub 2021 Nov 23. PMID 34816568
- [Result] Holtrop JS, Estabrooks PA, Gaglio B, Harden SM, Kessler RS, King DK, Kwan BM, Ory MG, Rabin BA, Shelton RC, Glasgow RE. Understanding and applying the RE-AIM framework: Clarifications and resources. J Clin Transl Sci. 2021 May 14;5(1):e126. doi: 10.1017/cts.2021.789. eCollection 2021. PMID 34367671
- [Result] Hegde S, Sreeram S, Bhat KR, Satish V, Shekar S, Babu M. Evaluation of post-COVID health status using the EuroQol-5D-5L scale. Pathog Glob Health. 2022 Dec;116(8):498-508. doi: 10.1080/20477724.2022.2035623. Epub 2022 Feb 7. PMID 35129097
- [Result] Guo J, Huang X, Dou L, Yan M, Shen T, Tang W, Li J. Aging and aging-related diseases: from molecular mechanisms to interventions and treatments. Signal Transduct Target Ther. 2022 Dec 16;7(1):391. doi: 10.1038/s41392-022-01251-0. PMID 36522308
- [Result] Guest, G., Bunce, A., & Johnson, L. (2006). How many interviews are enough? An experiment with data saturation and variability. Field methods, 18(1), 59-82.
- [Result] De Santis KK, Mergenthal L, Christianson L, Busskamp A, Vonstein C, Zeeb H. Digital Technologies for Health Promotion and Disease Prevention in Older People: Scoping Review. J Med Internet Res. 2023 Mar 23;25:e43542. doi: 10.2196/43542. PMID 36951896
- [Result] de Fatima Ribeiro Silva C, Ohara DG, Matos AP, Pinto ACPN, Pegorari MS. Short Physical Performance Battery as a Measure of Physical Performance and Mortality Predictor in Older Adults: A Comprehensive Literature Review. Int J Environ Res Public Health. 2021 Oct 10;18(20):10612. doi: 10.3390/ijerph182010612. PMID 34682359
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Result] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Result] Charlton K, Walton K, Brumerskyj K, Halcomb E, Hull A, Comerford T, do Rosario VA. Model of nutritional care in older adults: improving the identification and management of malnutrition using the Mini Nutritional Assessment–Short Form (MNA®-SF) in general practice. Aust J Prim Health. 2022 Feb;28(1):23-32. doi: 10.1071/PY21053. PMID 34911616
- [Result] Bahat G, Ozkok S, Kilic C, Karan MA. SARC-F Questionnaire Detects Frailty in Older Adults. J Nutr Health Aging. 2021;25(4):448-453. doi: 10.1007/s12603-020-1543-9. PMID 33786561